CLINICAL TRIAL: NCT07021963
Title: A Multicenter, Open-label Clinical Study to Evaluate the Long-term Safety of HRS-1893 in Hypertrophic Cardiomyopathy
Brief Title: A Clinical Study to Evaluate the Long-term Safety of HRS-1893 in Hypertrophic Cardiomyopathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1893-205
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obstructive Hypertrophic Cardiomyopathy Group (Experimental)
  Interventions: Drug: HRS-1893 Tablet
- Non-obstructive Hypertrophic Cardiomyopathy Group (Experimental)
  Interventions: Drug: HRS-1893 Tablet

INTERVENTIONS:
Drug: HRS-1893 Tablet — HRS-1893 tablet.

SUMMARY:
This study mainly evaluates the long-term safety of HRS-1893 in subjects with hypertrophic cardiomyopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with hypertrophic cardiomyopathy who have previously completed HRS-1893 related studies.
2. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose and must be non-lactating during the study. Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to refrain from donating sperm/eggs from the time they sign the informed consent form until 3 months after the last dose of trial drug, and to comply with relevant contraceptive requirements.
3. Understand the study procedures and methods, voluntarily participate in this trial, and sign the informed consent form in writing.

Exclusion Criteria:

1. Previous history of coronary artery disease (stenosis of one or more coronary arteries >70%) or myocardial infarction.
2. Have received medication for negative inotropic other than disopyramide, β-blocker, verapamil, diltiazem 4 weeks before screening.
3. History of syncope or sustained ventricular tachycardia within 6 months prior to screening.
4. Other conditions that the investigator considers the subject to be unsuitable for participating in this trial, such as physical or psychological diseases or conditions that may increase the risk of the trial, affect the subject's compliance with the protocol, or affect the subject's completion of the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs). | About 1 year.
Incidence of left ventricular ejection fraction (LVEF) <50%. | About 1 year.

SECONDARY OUTCOMES:
The change in cardiac troponin from baseline. | Week 24 and Week 52.
The change in N-terminal B-type natriuretic peptide (NT-proBNP) from baseline. | Week 24 and Week 52.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided